CLINICAL TRIAL: NCT04247737
Title: Effect of a Gluten Free Diet in Patients With IBS
Brief Title: Gluten Free Diet in IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, yurdagül zopf, Professor, University of Erlangen-Nürnberg Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IBS GFD
Record Dates: First submitted 2019-09-16; First posted 2020-01-30 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Gluten Sensitivity
Keywords: non-celiac glutensensitivity; irritable bowel syndrom
MeSH Terms: conditions — Celiac Disease | interventions — Diet, Gluten-Free

STUDY DESIGN:
Intervention Model Description: 25 healthy individuals and 150 patients with irritable bowel syndrome keep a gluten-free diet for six weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- gluten free diet (Experimental): six week gluten free diet
  Interventions: Other: gluten free diet

INTERVENTIONS:
Other: gluten free diet — Participants keep a gluten free diet for six weeks

SUMMARY:
Patients with irritable bowel syndrome (IBS) often benefit from dietary changes. The effect of a gluten-free diet (GFD) on clinical symptom improvement and psychological well-being will be checked in patients with IBS. In addition, the stimulatory potential of gluten on peripheral blood monocytes will be determined. Responders will be provoked with gluten containing bars or placebo bars to confirm the diagnosis of non-celiac glutensenstitivity.

DETAILED DESCRIPTION:
Patients with irritable bowel syndrome (IBS) often benefit from dietary changes. Since it has been shown that a gluten free diet (GFD) often alleviates the clinical symptoms, an overlap between patients with IBS and non-celiac glutensensitivity is assumed. The study includes 25 healthy individuals and 150 patients with IBS taking a six week GFD. Participants fill in questionnaires to determine clinical symptoms and psychological well being at the beginning and end of the dietary intervention. Patients with symptom relief under diet are further provoked in a double-blind placebo-controlled study with gluten or placebo containing bars for three weeks, separated by two weeks of washout to diagnosis of NCGS.

In addition, peripheral mononuclear cells are isolated at the beginning and end of the diet and the stimulating potential of wheat gluten is analyzed.

ELIGIBILITY:
Inclusion Criteria:

* healthy controls without gastrointestinal Symptoms
* patients with irritable bowel Syndrome (Rome IV criteria)

Exclusion Criteria:

* inflammatory bowel disease (Crohn's disease, Ulcerative colitis)
* celiac disease
* wheat allergy
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Determination of inflammatory Stimulation of monocytes after gluten exposure | six weeks
  Real-time PCR is used to determine the fold Change of gene expression of Interleukins IL-1ß and IL-6 after 24 hours of stimulation of peripheral monocytes with gluten Fragments (0,5 mg/ml)
Differences in Stimulation of inflammatory Parameters between healthy controls and patients with irritable bowel disease (IBD) | six weeks
  Detection of differences in relative gene Expression of inflammatory parameters (IL-1ß and IL-6) between patients with IBD and healthy controls

SECONDARY OUTCOMES:
Effect of a gluten free diet on improvement of gastrointestinal symptoms | six weeks
  Detection of patients with clinical improvement during gluten free diet, Determination of patients with at least >30% improvement in main gastrointestinal symptoms according the questionnaire for gastrointestinal symptomes (IBS-SSS)
Effect of the gluten free diet on Quality of life | six weeks
  Determination of the effect of a gluten free diet on Quality of Life using the Questionnaire psychological index for well being.
Determination of a subgroup of Patients with NCGS in IBS cohorte | six weeks
  Detection of patients with IBS that profite from a gluten free diet with Clinical improvement. Determination of the percentage of patients with NCGS compared to whole Population (n=150)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine 1, Hector Center for Nutrition, Exercise and Sports, Friedrich-Alexander-University Erlangen-Nuremberg, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No